CLINICAL TRIAL: NCT00673582
Title: Randomized, Multicentre, Double- Blind, Placebo Controlled Trial of Rosuvastatin 10 mg for Inhibition of Atherosclerosis Progression Assessed by Carotid Artery Ultrasound in HIV-positive Patients Treated With Antiretrovirals
Brief Title: Effectiveness of Rosuvastatin at Preventing the Progression of Atherosclerosis in HIV Positive Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor has withdrawn the funding
Sponsor: University of British Columbia (Other)
Collaborators: AstraZeneca (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Dr. Greg Bondy, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H07-00213; D3560L00059
Record Dates: First submitted 2008-04-30; First posted 2008-05-07 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Atherosclerosis; HIV Infections
Keywords: Statins; Intima Media Thickness; Plaque Area
MeSH Terms: conditions — Atherosclerosis; HIV Infections | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 10 mg/day rosuvastatin for 96 weeks
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg/day rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Placebo — Placebo, 10 mg a day for 96 weeks
  Arms: 2

SUMMARY:
Rosuvastatin is a drug used to lower cholesterol, which also has other cardiovascular benefits. The goal of this project is to determine if rosuvastatin is effective at slowing the development of heart disease in people with HIV. We expect that after 2 years of treatment people treated with rosuvastatin will show significantly better results than people treated with a placebo.

DETAILED DESCRIPTION:
HIV+ patients with at least one cardiovascular risk factor will be randomized to either rosuvastatin 10mg/day or placebo for a period of 96 weeks. B-mode carotid ultrasound will assess the primary outcome measure of average total thickness (a composite measurement of intima media thickness and total plaque area) at baseline, 24, 48, 72 and 96 weeks. We hypothesize that rosuvastatin will be significantly more effective with respect to inhibition of change in average total thickness between baseline and 96 weeks compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive, at least one cardiovascular disease risk factor

Exclusion Criteria:

* Diabetes
* Previous vascular disease
* Muscular disease
* Current use of other lipid lowering therapy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Average total thickness (a composite of carotid intima media thickness and total plaque area) | 96 weeks

SECONDARY OUTCOMES:
Carotid Intima Media Thickness, Total Plaque Area, Lipids | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greg Bondy, MD, Principal Investigator — University of British Columbia; Marianne Harris, MD, Study Director — University of British Columbia; Marek Smeija, MD, Study Director — University of British Columbia; Joel Singer, MD, Study Director — University of British Columbia; G.B. John Mancini, MD, Study Director — University of British Columbia; Sammy Chan, MD, Study Director — University of British Columbia; Julio Montaner, MD, Study Director — University of British Columbia
Locations (1):
- The St. Paul's Hospital HIV Metabolic Clinic & The BC Centre for Excellence in HIV/AIDS, Vancouver, British Columbia, Canada